## **INFORMED CONSENT FORM** to participate in:

## Effects of High-intensity Interval Circuit Training (HIICT) on the Cardiovascular and Functional Parameters of Aged Women

Ref: UALBIO2019/006

Date: 10/02/2019

## INFORMED CONSENT FORM. HIIT.

| FIRST NAME: |
|---|
| DNI: |
| Mr. Ismael Ballesta García, trainer of physical activity for elderly people, has duly informed, before th beginning of the session, about the main consequences that participants could suffer in performing session of high-intensity interval training, and the need of surpassing a previous recognition test prior th session. |
| Although the need of carrying out a prior recognition has been informed, the subject whose name and signature are shown below, insists on his wish to carry out the session, assuming, in case of occurrence, the possible pathological consequences. |
| Aim: Perform physical exercise at high heart rates. |
| Process: The participants could perform the following exercises: |
| 8 and 10 intervals work will be performed, depending on the demand of the activity, in which ratios of 2 of physical exercise will be carried out at low heart rates (Börg 10-11) and 1' at high heart rates (Börg 16). |
| The exercises consist in performing global movements in which large muscle groups are involved, at high speeds in the intervals of high-intensity and at low speed analytical movements in the low-intensity intervals. |
| Risks: May cause dizziness, falls, hypoglycemia and other causes discussed in the session. |
| Confidentiality: All personal data obtained is strictly confidential and will be analyzed anonymously. Only the research team and I will have access them and they'll be protected from any undue use: Ley 15/1999, de 13 diciembre. |
| Rights of the participant: At all times, I am free to stop collaborating if I desire so. There will be no sanctions or reprisals against m |
| I acknowledge that I participate freely under my own responsibility. I am aware of the information included in this form, I understand the procedures and I freely consent to perform the test and to take photographs while performing the session. |
| In , of 20 |
| Participant's Signature |